CLINICAL TRIAL: NCT04086368
Title: Derotational Femoral Osteotomy With Either Percutaneous Osteotomy and Intramedullary Nailing or Open Approach and Plating - a Randomized Controlled Trail
Brief Title: The FDR (Femoral Derotaton) Trail.
Acronym: FDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Grønseth, M.D. Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/2175
Record Dates: First submitted 2019-08-26; First posted 2019-09-11 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Increased Femoral Anteversion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Synthes Pediatric LCP Plate System (Active Comparator): Open osteotomy and osteofixation with the pediatric LCP hip plate
  Interventions: Device: Pediatric LCP Hip Plate System
- The adolescent Lateral Femoral Nail (Experimental): Percutaneous osteotomy and intramedullary nailing
  Interventions: Device: Adolescent Lateral Entry Femoral Nail

INTERVENTIONS:
Device: Adolescent Lateral Entry Femoral Nail — The use of an less invasive implant that has the same accuracy.
  Arms: The adolescent Lateral Femoral Nail
Device: Pediatric LCP Hip Plate System — Open approach to the femur where the osteotomy and osteofixation with plate and screws are preformed
  Arms: The Synthes Pediatric LCP Plate System

SUMMARY:
Femoral derotational osteotomy is the gold standard to correct symptomatic patients with increased femoral AV. There is no clear evidence in the literature supporting which surgical technique or implant that should be used. Traditionally these patients are treated with an open osteotomy and plate and screw fixation. In recent years intramedullary nailing with adolescent interlocking nail has been described and has shown to be a safe method. Percutaneous osteotomy and intramedullary nailing is considered a less invasive technique compared with open osteotomy and plate and screw fixation.

The primary objective of this project, is to investigate if derotational osteotomy by means of percutaneous osteotomy and nailing is a safe and accurate method compared to an open approach and plating.

DETAILED DESCRIPTION:
Introduction:

Gait deviations in children may be caused by excessive femoral anteversion (AV). This rotational deformity is usually self-limiting but is a common cause of parental concern. Femoral anteversion is an inward twisting (rotation) of the femur. Excessive femoral anteversion causes the patients knees and feet to turn inwards and have a "pigeon-toed" appearance. The AV angle can be measured in the transverse plane by a line through the centre of the femoral head and neck and a tangential line across of the posterior femoral condyles. In the majority of cases of increased femoral AV, normalization occurs spontaneously during growth.

Persisting excessive femoral torsion after the age of 8 years may lead to tripping and anterior hip and knee pain. Recent studies have shown that increased internal rotation is a risk factor for patellofemoral instability and may result in patellofemoral contact pressure.

There are no studies supporting conservative treatment with physiotherapy or braces. Femoral derotational osteotomy is the gold standard to correct symptomatic patients with increased femoral AV. Several techniques have been described and there is no clear evidence in the literature supporting which surgical technique or implant that should be used (3). Traditionally these patients are treated with an open osteotomy and plate and screw fixation. In recent years intramedullary nailing with adolescent interlocking nail has been described both for rotational osteotomies and femoral fractures. With a lateral trochanteric entry point this has been shown to be a safe method. Percutaneous osteotomy and intramedullary nailing is considered a less invasive technique compared with open osteotomy and plate and screw fixation.

Study aims:

The investigators want to compare percutaneous osteotomy and intramedullary nailing with an open approach and plating with interlocking screws, in a randomized, controlled single-center trial. Our hypothesis is that percutaneous osteotomy and intramedullary nailing is non-inferior in the treatment of increased femoral AV, compared to open approach with plate fixation.

The primary outcome measure is to measure the accuracy of the derotation at 12 months by CT scan.

Study design and methodology:

The study is a randomized non-inferiority trail comparing operative treatment of patients with symptomatic increased idiopathic femoral anteversion. There are two arms: (1) Open approach and plating and (2) percutaneous osteotomy and intramedullary nailing. The allocation ratio is 1:1.We will recruit patients in the age 10-18 years of age, referred to the Orthopedic department, Oslo University Hospital. A pediatric orthopedic surgeon will verify that the patient meets the inclusion criteria, and the patient will be given thorough oral and written information. After signed consent, the randomization allocation to treatment method will be performed by means of a web-solution made by NTNU WebCRF system with the approval from the OUS Head of Patient Security.

Follow-up:

The study patients will be followed-up over a one year period (6 weeks, 12 weeks, 12 months). All patients will be tested with 3 d gait analysis at 12 months and will be compared with the patients preoperativ 3 D gait analysis. All reoperations will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic findings: Femoral AV angle ≥ 30°
* Age 10-18 years.
* Hip or/and knee pain
* Less than 15 degrees external rotation of the hips

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria:

  * Previous femoral injury or illness which reduces the function of the extremity
  * Systemic or chronic injury or illness which reduces the function of the extremity
  * If the patient is not able to comply with study procedures

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2031-06-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the derotation | post operative (day1)
  Accuracy of the derotation measured in degrees on CT comparing the intended/planned correction with the actual derotation

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Children (KOOS-Child) | Baseline, 26 week and 52 week follow-up
  39 items divided in 5 subscales; Pain, other Symptoms (titled as "knee problems"), Difficulty during daily activities (ADL), Function in sport and play (Sport/Play) and Knee related Quality of Life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Visual analogue scale | Baseline, daily first six week. 4 times a day.
  General visual analog scale (VAS) for pain. scale is 0-10, where 10 is maximum pain og 0 is no pain. The scale is a 10 cm long line where the patient sets a mark. The actual level of pain is than measured on the scale from 0-10 (e.g. mark is at 5,5 cm - pain score 5,5)
KIDSCREEN-27 | Baseline, 26 week, 52 week follow-up
  The KIDSCREEN-27 is a globally used standardized health-related quality of life questionnaire measuring five Rasch scaled dimensions of wellbeing including: (1) Physical Well-being (5 items), (2) Psychological Well-being (7 items), (3) Autonomy and Parents (7 items), (4) Peers and Social Support (4 items), and (5) School Environment (4 items). Responses are indicated using a 5-point ordinal scale with responses ranging from 'never' to 'always', 'not at all' to 'extremely', or 'poor' to 'excellent'.

OTHER OUTCOMES:
Barnhöft | Baseline, 26 week, 52 week follow-up
  Six questions hip specific questionnaire regarding pain and function. Total score 0 - 100 points. 100 points describes no symptoms. Translated from the english version called The Children's Hospital Oakland Hip Evaluation Scale (CHOHES) - a modification of the Harris Hip Score.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grønseth, M.D, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway